CLINICAL TRIAL: NCT02220933
Title: Effect of MD1003 in Spinal Progressive Multiple Sclerosis: a Pivotal Randomized Double Blind Placebo Controlled Study
Brief Title: Effect of MD1003 in Spinal Progressive Multiple Sclerosis
Acronym: MS-SPI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD1003CT2013-02MS-SPI; 2013-002113-35 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; EDSS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MD1003 (Experimental): MD1003 100mg capsules, 1 capsule tid for 24 months
  Interventions: Drug: MD1003 100mg capsule
- Placebo (Placebo Comparator): Placebo capsule, 1 capsule tid for 12 months, then switch to MD1003 100mg capsule, 1 capsule tid for 12 months
  Interventions: Drug: MD1003 100mg capsule; Drug: Placebo

INTERVENTIONS:
Drug: MD1003 100mg capsule
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the superiority of MD1003 over placebo in the disability of patients suffering from progressive multiple sclerosis and especially those with gait impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis criteria of secondary or primary progressive MS with clinical evidence of spastic paraparesis fulfilling revised McDonald criteria (2010) and Lublin criteria (1996)
* Progression of the EDSS during the past two years of at least 1 point if EDSS from 4.5 to 5.5 and at least 0.5 point if EDSS from 6 to 7
* EDSS score from 4.5 to 7 (measured away from a relapse and confirmed at 6 months)
* Informed consent prior to any study procedure
* Patient aged 18-75 years

Exclusion Criteria:

* Any general chronic handicapping disease other than MS
* Intensive physical therapy program within the 3 months prior to inclusion
* Impossibility to perform the TW25 test
* New treatment introduced less than 3 months prior to inclusion or less than 1 month for Fampridine
* Pregnancy or woman with childbearing potential without contraception
* Evidence of inflammatory activity of the disease defined as "clinical evidence of a relapse during the year before inclusion or evidence of new gadolinium-enhanced lesions on a brain MRI performed the year before inclusion."

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients improved on either Expanded Disability Status Scale (EDSS) or time to walk 25 feet (TW25) | up to 24 months
  Proportions of patients in each treatment arm:
  - with decreased EDSS at M9 confirmed at Month12 (where decreased EDSS is defined as a decrease of at least 0.5 point if initial EDSS from 6 to 7 and a decrease of at least 1 point if initial EDSS from 4.5 to 5.5)
  or
  - with improved TW25 of at least 20% at Month 9 and Month12
  compared to the best EDSS and TW25 scores among screening visit (Month-1) and randomization visit (baseline)

SECONDARY OUTCOMES:
Multiple Sclerosis Walking Scale (MSWS) | Baseline, 12 months, 24 months
  The 12-item multiple sclerosis walking scale (MSWS-12) is a self-report measure of the impact of MS on the individual's walking ability.
Clinical Global Impression / Subject Global Impression (CGI / SGI) | 12 months, 24 months
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
  The clinical global impression will be assessed by the patient (subject global impression, SGI) and by the clinician (clinician global impression, CGI).
Unidimensional Fatigue Impact Scale (U-FIS) | Baseline, 12 months, 24 months
  The U-FIS has 22-items measuring the impact of fatigue.
Multiple Sclerosis Quality of Life Scale (SEP-59) | Baseline, 12 months, 24 months
  The SEP-59 is a multidimensional health-related quality of life measure that combines 36 generic items and 29 MS-specific items into a single instrument.
Hole Peg Test (9-HPT) | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
  The 9-HPT apparatus comprises a container with nine pegs and an empty pegboard with nine holes, set three by three. The pegs must be picked up one at a time and placed in the holes as quickly as possible until all holes are filled. Then, without pausing, the pegs should be removed one at a time, again as quickly as possible. This should be performed twice for each hand. If a peg falls onto the table, the peg should be picked up with the hand which is being tested. If a peg falls onto the floor, it is picked up by the examiner. The time is recorded in seconds, starting as the patient picks up the first peg and ending when the last peg drops into the container.

OTHER OUTCOMES:
Brain MRI | Baseline, 12 months
  Brain MRI using at least T2 and T1 sequences with gadolinium injection will be performed in a subset of 72 patients i.e 24 in the placebo group and 48 in the treated group, at study onset and after 12 months. Safety of MD1003 will be assessed by comparing novel T2 hypersignals as well as T1 post-gadolinium enhancing lesions in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Tourbah, MD, PhD, Principal Investigator — Hopital Maison Blanche, Reims, France; Frederic Sedel, MD, PhD, Study Director — Medday SAS, Paris, France
Locations (17):
- France (17):
  - Hopital Pellegrin, Bordeaux
  - Hopital de la cote de Nacre, Caen
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital general du Bocage, Dijon
  - Hopital Pierre Wertheimer, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - Hopital Central, Nancy
  - Hopital Nord Laennec, Nantes
  - Hopital Pasteur, Nice
  - Groupe hospitalier la Pitié-Salpêtrière, Paris
  - Fondation Rothschild, Paris
  - Centre hospitalier Intercommunal Poissy/Saint-Germain-en-Laye, Poissy
  - Hopital Maison Blanche, Reims
  - Hopital Pontchaillou, Rennes
  - Hopital Hautepierre, Strasbourg
  - Hopital Purpan, Toulouse